CLINICAL TRIAL: NCT06799884
Title: A Single-center, Open-label, Fixed-sequence Trial to Investigate the Effect of Multiple-dose Aprocitentan on the Single-dose Pharmacokinetics of Combined Oral Contraceptives in Healthy Female Participants
Brief Title: A Drug-drug Interaction Trial in Healthy Female Participants to Investigate the Effect of Aprocitentan on Combined Hormonal Contraceptives
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ID-080-111; 2024-517224-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-14; First posted 2025-01-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination; aprocitentan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ethinyl estradiol/levonorgestrel (LOETTE) (Experimental): In Trial Period A, participants will receive a single oral dose of 20µg ethinyl estradiol/100 µg levonorgestrel in the morning of Day 1.
  Interventions: Drug: Ethinyl Estradiol / Levonorgestrel Oral Tablet
- Aprocitentan (Experimental): In Trial Period B1, participants will receive a once daily oral dose of 25 mg aprocitentan in the morning of Day 1 to Day 9.
  Interventions: Drug: Aprocitentan
- Aprocitentan and ethinyl estradiol/levonorgestrel (LOETTE) (Experimental): In Trial Period B2, participants will receive a once daily oral dose of 25 mg aprocitentan in the morning of Day 10 to Day 13.
  On Day 10, participants will receive a single oral dose of 20µg ethinyl estradiol/100 µg levonorgestrel, administered concomitantly to aprocitentan.
  Interventions: Drug: Ethinyl Estradiol / Levonorgestrel Oral Tablet; Drug: Aprocitentan

INTERVENTIONS:
Drug: Ethinyl Estradiol / Levonorgestrel Oral Tablet — Coated tablet of 20 µg ethinyl estradiol and 100 µg levonorgestrel
  Other Names: LOETTE
  Arms: Aprocitentan and ethinyl estradiol/levonorgestrel (LOETTE); Ethinyl estradiol/levonorgestrel (LOETTE)
Drug: Aprocitentan — Film-coated tablet of aprocitentan 25 mg
  Arms: Aprocitentan; Aprocitentan and ethinyl estradiol/levonorgestrel (LOETTE)

SUMMARY:
The goal of this clinical trial is to learn if drug aprocitentan has an effect on hormonal contraceptives in healthy female volunteers. The main question it aims to answer is:

Does aprocitentan modify the fate of hormonal contraceptives in the body?

Trial participants will:

* Take a single dose of hormonal contraceptives (fixed combination) alone
* Take aprocitentan every day for 2 weeks
* Take a single dose of the same hormonal contraceptives at the same time as the 10th administration of aprocitentan.

DETAILED DESCRIPTION:
The main objective of the trial is to evaluate the influence of aprocitentan at steady-state on the single-dose pharmacokinetics (PK) of combined oral contraceptives.

19 healthy female participants will be enrolled to have at least 16 evaluable participants.

Following a screening period (from full signature of the informed consent form [ICF] to enrollment; 10 to 28 days prior to first trial intervention administration), eligible participants (meeting all inclusion criteria and none of the exclusion criteria) will be enrolled in the trial to participate in two sequential trial periods, Trial Period A and Trial Period B, with an in-between period of at least 7 days. Trial Period B will be split into two sequential sub-periods, Trial Period B1 and Trial Period B2.

* Trial Period A: Starts with a single administration of trial intervention on Day 1 and ends with an End-of-Trial Period (EoTP) assessment on Day 5. Trial intervention administration on Day 1 will be followed by a 96-hour observation period for safety monitoring and PK sampling.
* Trial Period B1: Trial intervention will be administered from Day 1 to Day 9, with assessments for PK sampling and safety monitoring performed throughout.
* Trial Period B2: Starts with administration of trial intervention on Day 10 and ends with an EoTP assessment on Day 14. Trial intervention will be administered from Day 10 to Day 13, with assessments for PK sampling and safety monitoring performed throughout.

Trial participation of an individual participant ends with the completion of the Participant Last Visit, which will be performed 10-14 days after the last administration of trial intervention. A post-trial safety follow up is performed 30-40 days after last administration of trial intervention.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form (ICF) prior to any trial-mandated procedure.
* Healthy female participants aged from 18 to 65 years at the time of signing the ICF.
* Ability to communicate well with the investigator, in a language understandable to the participant, and to understand and comply with the trial requirements.
* Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) at Screening.
* Normal or not clinically significant abnormal systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and pulse rate 45-90 bpm (inclusive), measured on either arm, after 5 min in the supine position at Screening and on Day 1 (predose) of Trial Period A (TP A).
* Participant of childbearing potential who has a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1 (predose) of TP A.
* Participant of childbearing potential who agrees to use two reliable methods of non- hormonal contraception from Screening and for at least 30 days after the last trial intervention administration, or be sexually inactive, or have a vasectomized partner.
* Participant of non-childbearing potential, i.e., postmenopausal (defined as 12 consecutive months with no menses without an alternative medical cause, confirmed by an follicle stimulating hormone test), with previous bilateral salpingectomy, bilateral salpingo-oophorectomy, or hysterectomy, or with premature ovarian failure (confirmed by a specialist), XY genotype, Turner syndrome, uterine agenesis).

Exclusion Criteria:

* Known hypersensitivity to aprocitentan, ethinylestradiol, or levonorgestrel, or treatments of the same class, or any of their excipients.
* Clinically relevant findings on the physical examination at Screening.
* Clinically relevant abnormalities on 12-lead electrocardiogram (ECG), measured after 5 min in a supine position at Screening or on Day 1 (pre-dose) of TP A.
* Clinically relevant findings in clinical laboratory tests (hematology and clinical chemistry) at Screening.
* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the trial interventions (appendectomy and herniotomy allowed if performed > 12 weeks prior to first trial intervention administration, cholecystectomy not allowed).
* Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation of the trial results.
* Previous clinically relevant history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Previous therapy with hormonal contraceptives or hormone replacement therapy within 2 months prior to first trial intervention administration.
* Pregnant, planning to become pregnant during the trial, or lactating participant of childbearing potential.
* Participant presenting any contraindications for LOETTE®

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of ethinyl estradiol/levonorgestrel | TP A: On Day 1 (pre-dose) and predefined times up to 96 hours post-dose (Day 5); TP B2: On Day 10 (pre-dose) and predefined times up to 96 hours post-dose (Day 14)
  The measured individual plasma concentrations will be used to directly obtain Cmax.
Time to maximum plasma concentration (tmax) of ethinyl estradiol/levonorgestrel | TP A: On Day 1 (pre-dose) and predefined times up to 96 hours post-dose (Day 5); TP B2: On Day 10 (pre-dose) and predefined times up to 96 hours post-dose (Day 14)
  The measured individual plasma concentrations will be used to directly obtain tmax.
Area under the Plasma Concentration-Time Curve (AUC 0-t) of ethinyl estradiol/levonorgestrel | TP A: On Day 1 (pre-dose) and predefined times up to 96 hours post-dose (Day 5); TP B2: On Day 10 (pre-dose) and predefined times up to 96 hours post-dose (Day 14)
  Change to AUC 0-t will be derived by non compartmental analysis of the concentration-time profiles.
Area under the Plasma Concentration-Time Curve (AUC 0-infinity) of ethinyl estradiol/levonorgestrel | TP A: On Day 1 (pre-dose) and predefined times up to 96 hours post-dose (Day 5); TP B2: On Day 10 (pre-dose) and predefined times up to 96 hours post-dose (Day 14)
  Change to AUC 0-infinity will be derived by non compartmental analysis of the concentration-time profiles.
Terminal half-life (t1/2) of ethinyl estradiol/levonorgestrel | TP A: On Day 1 (pre-dose) and predefined times up to 96 hours post-dose (Day 5); TP B2: On Day 10 (pre-dose) and predefined times up to 96 hours post-dose (Day 14)
  t1/2 will be derived by non compartmental analysis of the concentration-time profiles.
Trough plasma concentration (Ctrough) of aprocitentan | Prior to administration on Day 10, 11, 12 and 13 in TP B2
  Ctrough will be based on measured individual plasma concentrations of aprocitentan.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals
Locations (1):
- CEPHA s.r.o., Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No